CLINICAL TRIAL: NCT04053205
Title: An Multi-center, Open-label Phase Ib/II Study of Gentuximab Injection + Paclitaxel in Patients With Advanced Gastric or Gastroesophageal Junction Cancer to Evaluate Tolerability, Safety, Efficacy and Pharmacokinetics.
Brief Title: A Study of Gentuximab + Paclitaxel in Patients With Advanced Gastric or Gastroesophageal Junction Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai East Hospital (Other); Zhejiang University (Other); Fujian Tumor Hospital (Unknown); Sir Run Run Shaw Hospital (Other); The Affiliated Tumor Hospital of Harbin Medical University (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Tongji Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 043 CT
Record Dates: First submitted 2019-07-27; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Advanced Gastric or Gastroesophageal Junction Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 Gentuximab+ Paclitaxel (Experimental): 8 mg/kg Gentuximab administered intravenously (IV) on D1 and D15（28 days every cycle）+ 80 mg/m² paclitaxel administered IV on D1, D8 and D15
  Interventions: Drug: Gentuximab; Drug: Paclitaxel
- 2 Gentuximab+ Paclitaxel (Experimental): 12 mg/kg Gentuximab administered intravenously (IV) on D1 and D15（28 days every cycle）+ 80 mg/m² paclitaxel administered IV on D1, D8 and D15
  Interventions: Drug: Gentuximab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Gentuximab — Administered intravenously (IV)
Drug: Paclitaxel — Administered intravenously (IV)

SUMMARY:
The objective of the study is to evaluate Tolerability, Safety, and primary Efficacy of Gentuximab Injection at different dosage in combination with Paclitaxel in Advanced Gastric or Gastroesophageal Junction Cancer patients, to ensure adequate treatment dosage for further study. Meanwhile, the study also evaluate Pharmacokinetics of Gentuximab Injection at different dosage in combination with Paclitaxel.

DETAILED DESCRIPTION:
The study includes dose-limiting toxicity （DLT）observing period and randomization period with two cohorts as low-dose group（Gentuximab Injection 8mg/kg+ paclitaxel） and high-dose group（Gentuximab Injection 12mg/kg+ paclitaxel）. During the study，the anti-cancer efficacy, safety and anti-drug antibody were evaluated in all patients. DLT observation is only to subjects enrolled in DLT observation period and it lasts one treatment period. PK were doing in part of subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject can understand the process and methods of the study, complete the study in accordance with the protocol and is willing to sign a written informed consent.
* Male or female. aged between 18 and 75 years
* Histopathologically confirmed advanced advanced gastric or gastroesophageal junction cancer, and Documented progression during first-line fluoropyrimidine- and platinum- containing chemotherapy, or during the 3 months following the last cycle of such chemotherapy (or during the 6 months following the last dose of adjuvant therapy or new adjuvant therapy containing fluoropyrimidine and platinium).
* At least one Measurable lesion.
* ECOG Performance status (PS) score, 0-1 level.
* A life expectancy of >3 months.
* Adequate hematologic function, as defined by: Absolute neutrophil count (ANC) ≥1.5×109/L; hemoglobin concentration ≥90g/L (allowing blood transfusion); and platelet count ≥80×109/L.
* Adequate hepatic function, as defined by: ALT ≤ 2.5 × ULN, AST ≤ 2.5 × ULN, TBIL ≤ 1.5 × ULN (liver metastases patients ALT ≤ 5 × ULN, AST ≤ 5 × ULN, TBIL ≤ 3 × ULN).
* Adequate renal function, as defined by: serum creatinine level≤ 1.5 × ULN, or creatinine clearance ≥ 50ml / min when serum creatinine level> 1.5 × ULN.
* Adequate coagulation function, as defined by: International normalized ratio (INR) ≤1.5× ULN, activated partial thromboplastin time (aPTT) ≤1.5 x ULN.
* 24-hour urine protein quantitation is <1g（24-hour urine protein quantitative test should be performed when urine protein ≥1+ is found during screening visit）.
* Subjects (male and female) who have fertility must agree to use reliable contraceptive methods during the trial and in 3 months after the last administration. Female subjects in childbearing age must be negative for blood pregnancy test prior to enrollment.

Exclusion Criteria:

* Previously administrated with anti-angiogenic drugs or paclitaxel.
* Systematic anti-tumor therapy (non-anti-angiogenic drugs or paclitaxel) such as chemotherapy, radiotherapy, macromolecular targeted therapy, immunotherapy, endocrine therapy, etc. within 4 weeks before the first dose of investigational drug, except for the following: nitrourea or mitomycin C is within 6 weeks before the first dose, oral fluorouracil and small molecule targeted drugs are within 2 weeks or 5 half-life of the drug(whichever is longer) before the first dose，Chinese medicine with anti-cancer indications is within 2 weeks before the first dose.
* Has participated in a clinical study of a non-approved experimental agent within 4 weeks prior to screening visit.
* Has undergone major surgery within 4 weeks before screening visit (not including needle biopsy)， or would undergo planned surgery during the study.
* Subject with positive HCV-Ab, Anti-HIV or TP-Ab, or positive HBS-Ag with copies of HBV DNA > ULN.
* Patients with previously confirmed malignant tumors.
* History of arterial thrombosis or deep vein thrombosis within 6 months prior to screening, or a bleeding event no less than Grade level 3 within 2 months prior to screening， or the investigator determines that there is a risk of bleeding.
* History of severe cardiovascular and cerebrovascular diseases.
* Subjects with confirmed brain tumor metastases，but subjects in steady situation can be enrolled.
* Active bleeding confirmed by gastroscopy when fecal occult blood positive (only subjects with primary lesions not removed need to do fecal occult blood test.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 12 months before screening visit.
* Thoracic，abdominal or pericardial effusion that cannot be controlled by repeated drainage or with obvious symptoms.
* Has a nonhealing wound, serious ulcer, or unrecovered bone fracture.
* Active infections requiring systemic treatment, including but not limited to active tuberculosis.
* Using anticoagulation and antiplatelet drugs.
* Female subjects who is pregnant (confirmed by urine or serum pregnancy test) or lactating.
* Has a known serious allergy reaction to recombination monoclonal antibody (MAb) drug, ,or infusion reaction.
* Has known alcohol or drug dependency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | Up to 4 Weeks
  Number of Participants With One or More Drug-Related Adverse Events (AEs) defined as DLT in the protocol
AEs or SAEs | Baseline through Study Completion, about 24 weeks
  Drug-Related Adverse Events (AEs) or Any Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Objective response rate（ORR） | Up to 6 cycles (28 days for every cycle)
  Proportion of Participants With CR and PR
Progression-free survival (PFS) | Up to 6 cycles (28 days for every cycle)
  The time from randomization to the patient tumor progression or death.
Disease control rate (DCR) | Up to 6 cycles (28 days for every cycle)
  Proportion of Participants With CR, PR and SD
Time-to-progress (TTP) | Up to 6 cycles (28 days for every cycle)
  The time from randomization to the patient tumor progression.
Time-to-failure (TTF) | Up to 6 cycles (28 days for every cycle)
  The time from randomization to the patient withdraw from the study.
Anti-drug antibody | Up to 6 cycles (28 days for every cycle)
  Number of Participants With Anti-drug Antibodies
Pharmacokinetics Cmax | Cycle 1(day1-day 15)& Cycle 2(day 15-day26) & Cycle 3(day 1) (28 days for every cycle)
  Maximum Concentration (Cmax)
Area Under the Concentration-Time Curve (AUC) | Cycle 1(day1-day 15)& Cycle 2(day 15-day26) & Cycle 3(day 1) Cycle 1(day1-day 15)& Cycle 2(day 15-day26) & Cycle 3(day 1) （28 days for every cycle）

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Fujian Tumor Hospital, Fuzhou, Fujian
  - The Sixth Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Hangzhou, Zhejiang
  - Shanghai East Hospital, Shanghai
  - Shanghai First People's Hospital, Shanghai